CLINICAL TRIAL: NCT00772603
Title: Phase III Study to Evaluate the Efficacy and Safety of OXC XR as Adjunctive Therapy in Subjects With Refractory Partial Seizures
Brief Title: Evaluation of Efficacy and Safety of OXC XR as Adjunctive Therapy for Partial Seizures
Acronym: PROSPER1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 804P301
Record Dates: First submitted 2008-10-10; First posted 2008-10-15 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-12

CONDITIONS: Epilepsies, Partial
Keywords: Partial onset epilepsy; Partial onset seizures
MeSH Terms: conditions — Epilepsies, Partial | interventions — Oxcarbazepine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo - four identical tablets taken orally once daily
  Interventions: Drug: Placebo
- 2400 mg SPN-804 (Active Comparator): 2400mg OXC XR taken orally once daily as four identical tablets
  Interventions: Drug: 2400mg SPN-804
- 1200mg SPN-804 (Active Comparator): 1200mg OXC XR taken orally once daily as four identical tablets
  Interventions: Drug: 1200mg SPN-804

INTERVENTIONS:
Drug: Placebo — Non-active tablet identical to study drug tablets
  Other Names: sham treatment
  Arms: Placebo
Drug: 2400mg SPN-804 — tablets containing 600mg OXC XR, identical to non-active tablets
  Other Names: Oxcarbazepine extended-release; Oxtellar XR; Oxtellar
  Arms: 2400 mg SPN-804
Drug: 1200mg SPN-804 — two active tablets and two non-active tablets, all identical
  Other Names: Oxcarbazepine extended-release; Oxtellar XR; Oxtellar
  Arms: 1200mg SPN-804

SUMMARY:
Evaluation of the safety and efficacy of Oxcarbazepine XR as adjunctive treatment for adults with partial onset seizures

DETAILED DESCRIPTION:
Multicenter, double-blind, randomized, placebo-controlled, three-arm. parallel-group study of the efficacy and safety of extended-release oxcarbazepine in the treatment of adults with refractory partial onset epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Capable of complying with the study procedures.
* Able to provide written informed consent
* Male or female aged 18 to 65 years, inclusive.
* Diagnosis of partial onset seizures
* Minimum of three seizures per 28 days
* Receiving treatment with 1-3 AEDs
* Refractory to at least one AED
* No progressive neurological conditions by recent MRI/CT
* Adequate birth control in women of child-bearing potential

Exclusion Criteria:

* Refractory to OXC for reasons of efficacy
* Recent status epilepticus
* Recent non-epileptic seizures
* Current diagnosis of major depression
* Recent suicidal plan or intent or more than one attempt
* Current use of oxcarbazepine, felbamate for < 18 months, phenytoin with levels >15mcg/mL or frequent need for rescue benzodiazepines
* Current use of sodium-lowering non-seizure medications.
* Clinically significant hepatic, renal, or cardiovascular function
* History of recent substance abuse
* Females who are pregnant or lactating.
* Hypersensitivity to OXC or related drugs
* Difficulty swallowing study medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet K Johnson, PhD, Study Director — Supernus Pharmaceuticals, Inc.
Locations (71):
- United States (23):
  - Huntsville, Alabama
  - Northport, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Riverside, California
  - West Los Angeles, California
  - Aurora, Colorado
  - Jacksonville, Florida
  - Miami, Florida
  - Sarasota, Florida
  - Atlanta, Georgia
  - Springfield, Illinois
  - Lexington, Kentucky
  - Bethesda, Maryland
  - Missoula, Montana
  - Camden, New Jersey
  - New York, New York
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Baytown, Texas
  - Temple, Texas
- Bulgaria (6):
  - Blagoevgrad
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Varna
- Canada (2):
  - Edmonton, Alberta
  - Greenfield Park, Quebec
- Croatia (4):
  - Dubrovnik
  - Rijeka
  - Zadar
  - Zagreb
- Mexico (11):
  - Aguascalientes, Aguascalientes
  - Chihuahua City, Chihuahua
  - Ciudad Juárez, Chihuahua
  - Durango, Durango
  - Guadalajara, Jalisco
  - Zapopan, Jalisco
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - Puebla City, Puebla
  - San Luis Potosí City, San Luis Potosí
  - Toluca, State of Mexico
- Poland (9):
  - Giżycko
  - Gmina Końskie
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Warsaw
  - Wilkowice
  - Zabrze
- Romania (4):
  - Bucharest
  - Campulung Muscel
  - Cluj-Napoca
  - Craiova
- Russia (12):
  - Saint Petersburg, Sestroretsk
  - Kazan'
  - Kirov
  - Kursk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Pyatigorsk
  - Saint Petersburg
  - Samara
  - Smolensk
  - Yaroslavl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients with refractory partial onset epilepsy were recruited from December 2009 to March 2011 at clinical sites in 8 countries.
Pre-assignment Details: Patients had at least three partial seizures per 28 days during an 8 week Baseline Period. Subjects were receiving treatment with one to three antiepileptic drugs and were on stable treatment for a minimum of 4 weeks. Subjects with a diagnosis other than partial epilepsy were excluded.
Groups:
- 2400mg/Day SPN-804: 2400mg of SPN-804O once daily
- 1200mg/Day SPN-804: 1200mg SPN-804O once daily
- Placebo: Placebo once daily
Period: Overall Study
Arm/Group | 2400mg/Day SPN-804 | 1200mg/Day SPN-804 | Placebo
Started | 123 | 122 | 121
Completed | 71 | 82 | 95
Not Completed | 52 | 40 | 26
Not completed — Withdrawal by Subject | 11 | 10 | 6
Not completed — Adverse Event | 37 | 18 | 10
Not completed — Subject Non-compliance | 1 | 6 | 4
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 5 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Other | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- 2400mg/Day SPN-804: 2400mg SPN-804O once daily
- 1200mg/Day SPN-804: 1200mg SPN-804O given once daily
- Placebo: Placebo given once daily.
- Total: Total of all reporting groups
Arm/Group | 2400mg/Day SPN-804 | 1200mg/Day SPN-804 | Placebo | Total
Number analyzed (Participants) | 123 | 122 | 121 | 366
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 123 | 122 | 121 | 366
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (11.58) | 39.1 (11.51) | 39.1 (12.49) | 38.9 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 71 | 67 | 202
  Male | 59 | 51 | 54 | 164
Region of Enrollment [Number; unit: participants]
  United States | 20 | 23 | 26 | 69
  Mexico | 15 | 16 | 14 | 45
  Canada | 0 | 1 | 1 | 2
  Poland | 25 | 16 | 13 | 54
  Romania | 8 | 10 | 6 | 24
  Croatia | 10 | 7 | 12 | 29
  Russian Federation | 28 | 31 | 31 | 90
  Bulgaria | 17 | 18 | 18 | 53

OUTCOME MEASURES:

1. Primary Outcome: PCH(T), ITT
Description: Percent change (PCH) in seizure frequency per 28d relative to Baseline, Treatment Phase (PCH[T]), Intent-to-Treat population.
Time Frame: Change at 16 weeks (4wks Titration + 12 wks Maintenance) compared to Baseline
Population: All safety population subjects with baseline Seizure Diary data and at least one visit during the Treatment Phase (ITT population). Subjects must have had at least 3 consecutive weeks of Seizure Diary data (SDD) in the Baseline Phase and at least 14 consecutive days of SDD after starting study drug.
Measure: Median (Full Range); unit: percentage of change
Groups:
- 2400mg/Day SPN-804: 2400mg SPN-804 once daily
- 1200mg/Day SPN-804: 1200mg SPN-804 once daily
Arm/Group | 2400mg/Day SPN-804 | 1200mg/Day SPN-804 | Placebo
Number analyzed (Participants) | 111 | 109 | 117
percentage of change | -42.90 (53.11) [-100.0 to 212.8] | -38.20 (69.84) [-100.0 to 556.1] | -28.70 (67.34) [-100.0 to 333.6]
Statistical Analysis 1: Comparison: 2400mg/Day SPN-804 vs Placebo; A Wilcoxon rank-sum test was used to test the hypothesis of equal median reduction in PCH(T) from baseline between SPN-804 and placebo. The sample size of 120 patients per treatment arm provides over 95% power to detect a difference of 31% to 42% between placebo and 2400mg SPN-804 at a two-sided 0.025 level for an overall Type I error rate of 0.050; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney) — P values reported are not adjusted for multiple comparisons. To preserve the overall Type I error-rate at 0.050, a step-up Hochberg procedure was used for the pair-wise comparisons; Median Difference (Net) = -18.30, 95% CI 2-sided [-30.40 to -5.80]
Statistical Analysis 2: Comparison: 1200mg/Day SPN-804 vs Placebo; A Wilcoxon rank-sum test was used to test the hypothesis of equal median reduction in PCH(T) from baseline between SPN-804 and placebo. The sample size of 120 patients per treatment arm provides over 95% power to detect a difference of 24% to 32% between placebo and 1200mg SPN-804 at a two-sided 0.025 level for an overall Type I error rate of 0.050; Test type: Superiority or Other; p = 0.078, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]; Median Difference (Net) = -10.30, 95% CI 2-sided [-22.30 to 1.20]

2. Secondary Outcome: PCH(M)- ITT
Description: Percent change in seizure frequency per 28 days relative to Baseline, Maintenance Period (PCH[M]), Intent-to-Treat population
Time Frame: Change at 12 weeks (Maintenance Period) compared to Baseline
Population: All safety population subjects with adequate baseline Seizure Diary data (at least three consecutive weeks) and at least one visit during the Titration Period and one visit during the Maintenance Period.
Measure: Median (95% Confidence Interval); unit: percentage of change
Arm/Group | 2400mg/Day SPN-804 | 1200mg/Day SPN-804 | Placebo
Number analyzed (Participants) | 88 | 97 | 109
percentage of change | -49.15 [-100 to 158] | -35.30 [-100 to 690.5] | -32.90 [-100 to 212.6]
Statistical Analysis 1: Comparison: 2400mg/Day SPN-804 vs Placebo; A Wilcoxon rank-sum test was used to test the hypothesis of equal median reduction in PCH(M) from baseline between SPN-804 and placebo. The sample size of 120 patients per treatment arm provides over 95% power to detect a difference of 31% to 42% between placebo and 2400mg SPN-804 at a two-sided 0.025 level for an overall Type I error rate of 0.050; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]; Median Difference (Net) = -33.00, 95% CI 2-sided [-33.00 to -6.30]
Statistical Analysis 2: Comparison: 1200mg/Day SPN-804 vs Placebo; A Wilcoxon rank-sum test was used to test the hypothesis of equal median reduction in PCH(M) from baseline between SPN-804 and placebo. The sample size of 120 patients per treatment arm provides over 95% power to detect a difference of 24% to 32% between placebo and 1200mg SPN-804 at a two-sided 0.025 level for an overall Type I error rate of 0.050; Test type: Superiority or Other; p = 0.589, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]; Median Difference (Net) = -3.30, 95% CI 2-sided [-16.20 to 9.70]

3. Secondary Outcome: Responder Rate, ITT
Description: Percent of patients with a positive response, defined as a 50% or greater reduction in seizure frequency per 28 days relative to Baseline, Treatment Phase, Intent-to-Treat population
Time Frame: At the end of 16 weeks (4 wks Titration + 12 wks Maintenance)
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | 2400mg/Day SPN-804 | 1200mg/Day SPN-804 | Placebo
Number analyzed (Participants) | 109 | 111 | 117
percentage of patients | 50 | 44 | 34
Statistical Analysis 1: Comparison: 2400mg/Day SPN-804 vs Placebo; The treatment response was analyzed using a logistic regression model with treatment group as a factor and country (or cluster), age, sex, and baseline seizure frequency per 28 days as explanatory variables; Test type: Superiority or Other; p = 0.018, Regression, Logistic; Odds Ratio (OR) = 1.983, 95% CI 2-sided [1.126 to 3.494]
Statistical Analysis 2: Comparison: 1200mg/Day SPN-804 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.075, Regression, Logistic; Odds Ratio (OR) = 1.670, 95% CI [0.950 to 2.937]

4. Secondary Outcome: Seizure-Free Rates, ITT
Description: Percent of patients seizure-free during Treatment Phase, Intent-to-Treat population
Time Frame: At the end of 16 weeks (4 wks Titration + 12 wks Maintenance)
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | 2400mg/Day SPN-804 | 1200mg/Day SPN-804 | Placebo
Number analyzed (Participants) | 111 | 109 | 117
percentage of patients | 14 | 6 | 4
Statistical Analysis 1: Comparison: 2400mg/Day SPN-804 vs Placebo; Pairwise comparisons of OXC XR 2400mg/day vs. placebo seizure-free rates during the Treatment Phase were made by means of Fisher's exact test for the ITT population; Test type: Superiority or Other; p = 0.013, Fisher Exact
Statistical Analysis 2: Comparison: 1200mg/Day SPN-804 vs Placebo; Pairwise comparisons of OXC XR 1200mg/day vs. placebo seizure-free rates during the Treatment Phase were made by means of Fisher's exact test for the ITT population; Test type: Superiority or Other; p = 0.528, Fisher Exact

5. Secondary Outcome: Seizure Free Rate, ITT, (M)
Description: Percent of patients seizure-free during Maintenance, Intent-to-Treat population
Time Frame: At the end of 12 weeks (Maintenance Period)
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | 2400mg/Day SPN-804 | 1200mg/Day SPN-804 | Placebo
Number analyzed (Participants) | 88 | 97 | 109
percentage of patients | 17 | 4 | 7
Statistical Analysis 1: Comparison: 2400mg/Day SPN-804 vs Placebo; Pairwise comparisons of OXC XR 2400mg/day vs. placebo seizure-free rates during the Maintenance Period were made by means of Fisher's exact test for the ITT population; Test type: Superiority or Other; p = 0.008, Fisher Exact
Statistical Analysis 2: Comparison: 1200mg/Day SPN-804 vs Placebo; Pairwise comparisons of OXC XR 1200mg/day vs. placebo seizure-free rates during the Maintenance Period were made by means of Fisher's exact test for the ITT population; Test type: Superiority or Other; p = 0.0546, Fisher Exact

ADVERSE EVENTS:
Time Frame: All randomized subjects who took at least one dose of study drug.
Description: Safety was assessed using adverse events (AEs), clinical laboratory results, vital signs, physical and neurological examinations, and electrocardiograms (ECGs).
Groups:
- 2400mg/Day SPN-804: 2400mg total daily dose of SPN-804O once a day (QD), given as four 600mg tablets
- 1200mg/Day SPN-804: 1200mg total daily dose of SPN-804O QD, given as two 600mg tablets and two identical placebo tablets.
- Placebo: placebo QD, given as four placebo tablets
Arm/Group | 2400mg/Day SPN-804 | 1200mg/Day SPN-804 | Placebo
Serious Adverse Events (participants affected / at risk) | 10/123 | 7/122 | 7/121
Other Adverse Events (participants affected / at risk) | 69/123 | 57/122 | 55/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2400mg/Day SPN-804 (N=123) | 1200mg/Day SPN-804 (N=122) | Placebo (N=121)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Drug intolerance (General disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skull fractured, base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatreamia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Pituitary tumor, benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Convulsions/complex partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Post-ictal state (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2400mg/Day SPN-804 (N=123) | 1200mg/Day SPN-804 (N=122) | Placebo (N=121)
Dizziness (Nervous system disorders) | 50 (60) | 24 (30) | 18 (21)
Somnolence (Nervous system disorders) | 17 (19) | 14 (14) | 11 (12)
Headache (Nervous system disorders) | 19 (21) | 10 (10) | 9 (12)
Balance Disorder (Nervous system disorders) | 8 (12) | 6 (11) | 6 (7)
Vomiting (Gastrointestinal disorders) | 19 (20) | 7 (10) | 11 (11)
Diplopia (Eye disorders) | 16 (21) | 12 (15) | 5 (5)
Asthenia (General disorders) | 9 (9) | 4 (4) | 1 (2)
Fatigue (General disorders) | 4 (5) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other